CLINICAL TRIAL: NCT06047678
Title: Acute Effect of Individual Variants of Agonist-antagonist and Traditional Agonistic Resistance Training on Cardiovascular Parameters in Patients With Normotension and 1 Stage of Hypertension.
Brief Title: Acute Effect of Individual Variants of Agonist-antagonist and Traditional Agonistic Resistance Training on Cardiovascular Parameters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Roman Jurik, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CharlesUCRFTVS
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Arterial Stiffness; Hypertension; Cardiovascular Diseases
Keywords: resistance training; arterial stiffness; hypertension; cardiovascular health
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Comparing two groups
  1. Normotensive group
  2. Hypertension Stage 1 group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normotension group (Experimental): Participants with normotension Adult: 40 - 63 years old Physically active - no professional sportsman
  Interventions: Behavioral: Cardiovascular fitness
- Hypertension Stage 1 group (Experimental): Participants with Hypertension Stage 1 Adult: 40 - 63 years old Physically active - no professional sportsman.
  Interventions: Behavioral: Cardiovascular fitness

INTERVENTIONS:
Behavioral: Cardiovascular fitness — A randomized single-blind controlled trial tested the hypothesis that different variants of resistance training (antagonistic lower and upper body training, agonistic lower and upper body training, and aerobic training) have different effects on blood pressure (systolic and diastolic), aortic pulse wave velocity (PWVao), and augmentation index (Aix) values and compared subjects with normotension and hypertension during and after exercise session.

SUMMARY:
Prevention and non pharmacological treatment of prehypertension and hypertension stage 1

The effect of individual variants of agonist-antagonist and traditional agonistic resistance training on cardiovascular parameters in individuals with normotension and hypertension.

What does the study involve?

1. Cardiovascular parameters
2. Body composition
3. Blood tests for heart disease
4. Training intervention

A. Resistance training protocol: 75% 1RM, 10 reps, 3 sets, 2 min rest between sets and exercises, 16 exercises

1. Agonistic RT - upper body
2. Agonistic RT - lower body
3. Agonist-Antagonist - upper body
4. Agonist-Antagonist - lower body B. Aerobic training: 60% SF max, 4 x 10 min, 2 min rest between sets
5. Intraabdominal wall tension activity
6. The Borg rating of perceived exertion
7. Handgrip testing
8. Repetition testing (RM)

DETAILED DESCRIPTION:
The effect of individual variants of agonist-antagonist and traditional agonistic resistance training on cardiovascular parameters in individuals with normotension and hypertension.

Participants with normotension and hypertension (1 stage of hypertension), adult: 40 - 63 years old, physically active - no professional sportsman.

Participants with fluctuating blood pressure, with type 1 and type 2 diabetes mellitus, after a myocardial infarction, after a stroke, with an infectious disease, with grade 3 obesity, with hypertension II. - IV. degrees and individuals suffering from dizziness during exercise are excluded.

What does the study involve?

1. Cardiovascular parameters - SBP, DBP, HR, PWV and augmentation index are measure by Arteriograph (TensioMed, Budapest, Hungary) at baseline, during and after training sessions.
2. Body composition - Body composition is measured by InBody370S in Pavel Kolar´s Centre of Physical Medicine before intervention.
3. Blood tests for heart disease - tests help determine the risk of heart diseases. it can be very helpful in assessing health. Total cholesterol, LDL, HDL, triacylglycerols, CRP, glucose are measured by NEXTCLINICS Czech a.s. before intervention
4. Training intervention: Resistance training: 75% 1RM, 10 reps, 3 sets, 2 min rest between sets and exercises, 16 exercises (8 lower body exercise + 8 upper body exercise), Agonistic vs Agonistic-antagonist resistance training, freeweight + cable machines according to ACSM's Guidelines for Exercise Testing and Prescription, 11th Edition

A. Resistance training protocol:

1. Agonistic RT - upper body
2. Agonistic RT - lower body
3. Agonist-Antagonist - upper body
4. Agonist-Antagonist - lower body B. Aerobic training: 60% SF max, 4 x 10 min, 2 min rest between sets
5. Intraabdominal wall tension testing during resistance training - correction of respiratory stereotype during exercise. Abdominal wall tension is measured by OHMBelt (Nilus Medical LLC) in Pavel Kolar´s Centre of Physical Medicine before, during and after resistance training.
6. The intensity of the exercises is determined by the Borg rating of perceived exertion (RPE) during resistance training.
7. Handgrip is measured by Takei (TKK 5401, Japan) before intervention. The Harvard Step Test is used to measure a clients aerobic fitness before intervention.
8. Repetition testing is assessing the strength capacity of individuals in non-laboratory environments: 15 RM, 10RM, 5 RM, 1 RM tests in Pavel Kolar´s Centre of Physical Medicine and the Faculty of Physical Education and Sport, Charles University before intervention.

Benefits: health assessment, physical fitness testing, professional supervision of training.

Potential disadvantages: soreness and muscle strain, fatigue, dizziness, feeling sick.

The study is run in Pavel Kolar´s Centre of Physical Medicine and the Faculty of Physical Education and Sport, Charles University.

The study began in April 2022 and will run until December 31, 2023. Agonist-Antagonist resistance training with 75% 1 RM induces an similar decrease in systolic and diastolic blood pressure values after training sessions at the p<0.05 level, as aerobic (control) training in normotensive and hypertensive individuals (1 stage of hypertension).

Alternative hypothesis H1: Agonistic-Antagonist resistance training with 75% 1 RM will result in a smaller increase in systolic and diastolic blood pressure values after training sessions at the p<0.05 level, compared to traditional resistance training in sets in normotensive and hypertensive subjects (1 stage of hypertension).

Agonistic resistance training with 75% 1 RM will induce a similar increase in pulse wave velocity during the training sessions at the p <0.05 level as aerobic (control) training in normotensive and hypertensive subjects (1 stage of hypertension).

Alternative Hypothesis H2: Agonistic resistance training with 75% 1 RM will result in a statistically significantly greater increase in pulse wave velocity values during the training sessions at the p <0.05 level compared to traditional resistance training in sets in normotensive and hypertensive subjects (1 stage of hypertension).

Isolated exercises induce a similar increase in systolic and diastolic blood pressure values during resistance training in normotensive and hypertensive individuals (1 stage of hypertension) as aerobic (control) training.

Alternative hypothesis H3: Complex/multi-joint exercises will lead to statistically significantly higher increases in systolic and diastolic blood pressure values in normotensive and hypertensive subjects (1 stage of hypertension) compared to isolated exercises.

ELIGIBILITY:
Inclusion Criteria:

* participants with normotension and clinical diagnosis of hypertension (1 stage of hypertension)
* adult: 40 - 63 years old
* physically active
* capable of strength and aerobic training

Exclusion Criteria:

* fluctuating blood pressure
* type 1 and type 2 diabetes mellitus
* after a myocardial infarction
* after a stroke
* with an infectious disease
* with grade 3 obesity
* hypertension II. - IV. degrees
* suffering from dizziness during exercise

Ages: 40 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness - Pulse wave velocity | The training takes place twice a week, 1 training session takes 60 minutes, the total number of sessions is 5. The total length of the program is 3 weeks, duration is 5 hours.
  Specifically, Aortic pulse wave velocity will be measured. The norm is up to 9 m/s, values above 9 m/s indicate impaired arterial stiffness. Arterial stiffness is a growing epidemic associated with increased risk of cardiovascular events, dementia, and death. Decreased compliance of the central vasculature alters arterial pressure and flow dynamics and impacts cardiac performance and coronary perfusion. It is measured by Arteriograph (TensioMed, Budapest, Hungary).
Blood pressure | The training takes place twice a week, 1 training session takes 60 minutes, the total number of sessions is 5. The total length of the program is 3 weeks, duration is 5 hours.
  Measurement of changes in blood pressure level. Increase in systolic and diastolic blood pressure (mm Hg) during resistance training for agonist-antagonist and traditional agonist resistance training. Blood pressure ranges:
  Normal: less than 120 systolic and 80 diastolic. Elevated: 120-129 systolic and less than 80 diastolic. Stage 1 hypertension: 130-139 systolic or 80-89 diastolic. Stage 2 hypertension: at least 140 systolic or at least 90 diastolic.Investigators are looking for the safest option of resistance training for individuals with hypertension. It is measured by Arteriograph (TensioMed, Budapest, Hungary).

SECONDARY OUTCOMES:
Handgrip strength | before intervention, one session, it takes 10 minutes, week 1
  Handgrip (kg) is measured by Takei (TKK 5401, Japan).It will be measured for both hands (left and right). Three trials will be performed on each hand and the mean will be calculated. The standard for men over 40 years of age is 47 (±9.5) kg for the right hand and 45 (±9.3) kg for the left hand. The standard for women over 40 is 29 (±5.7) kg for the right hand and 28 (±5.7) kg for the left hand. Higher values are considered to be better.
The concentration of total cholesterol | before intervention, one session, it takes 15 minutes, week 1
  Total cholestero (mmol/l) is measured by NEXTCLINICS Czech a.s. The reference range is 2,90-5,00 mmol/l.
Body mass index | before intervention, one session, it takes 15 minutes, week 1
  BMI (kg/m2 ) is measured by InBody370S. Optimal values for BMI: 18.5-24.9 kg
Harvard step test | before intervention, one session, it takes 8 minutes, week 1
  The Harvard Step Test is used to measure a clients aerobic fitness, being a predictive test of their VO2max. It tests the cardiovascular system and reflects the general capacity of body to cope with increased physical work load and ability to recover from it. Values in steptest for untrained population: > 90 points: excellent, 80-89 points: good, < 65 - 79 points: average, 55 - 64 points: Poor, 65 - 79: low average. Higher values mean a better result.
Abdominal wall tension | two measurements, 2x 60-90 minutes, week 1
  Abdominal wall tension is measured by OHMBelt (Nilus Medical LLC) . Increases in abdominal wall tension correlate with intra-abdominal pressure changes. It could be an approximate predictor of systolic blood pressure.
The Borg rating of perceived exertion | The total length of the program is 3 weeks, total duration is 5 hours. The results are recorded after each series of exercises - total 8x
  A modified Borg CR10 Scale will be used in this study. The subject will indicate the intensity of the exercise on a scale from 0 to 10. 0 means no exertion and 10 means maximum exertion.
Repetition testing | two measurements, 2x 60-90 minutes, week 1
  Assessing the strength capacity of individuals in non-laboratory environments. It is simply defined as the maximal or submacimal weight an individual can lift for only one repetition with correct technique. We measured 15 RM, 10 RM, 5 RM, 5 RM and 1RM in normotensive individuals.
Fat mass | before intervention, one session, it takes 15 minutes, week 1
  Fat mass (kg) is measured by InBody370S.
Lean mass | before intervention, one session, it takes 15 minutes, week 1
  Lean mass (kg) is measured by InBody370S.
Body fat | before intervention, one session, it takes 15 minutes, week 1
  Body fat (%) is measured by InBody370S. Optimal values for % body fat: age 40-59 - 23-33% body fat, age 60-79 - 24-35% body fat.
Body weight | before intervention, one session, it takes 15 minutes, week 1
  Body weight (kg) is measured by InBody370S.
The concentration of low density lipoprotein (LDL) | before intervention, one session, it takes 15 minutes, week 1
  LDL (mmol/l) is measured by NEXTCLINICS Czech a.s. The reference range is 1,2-3,00 mmol/l.
The concentration of high density lipoprotein (HDL) | before intervention, one session, it takes 15 minutes, week 1
  HDL (mmol/l) is measured by NEXTCLINICS Czech a.s. The reference range is 1,00-2,10 mmol/l.
The concentration of triacylglycerols | before intervention, one session, it takes 15 minutes, week 1
  Triacylglycerols (mmol/l) are measured by NEXTCLINICS Czech a.s. The reference range is 0,45-1,70 mmol/l.
The concentration of c-reactive protein (CRP) | before intervention, one session, it takes 15 minutes, week 1
  CRP (mg/l) is measured by NEXTCLINICS Czech a.s. The reference range is 0,0-8,0 mmol/l.
Blood sugar level | before intervention, one session, it takes 15 minutes, week 1
  Blood sugar (mmol/l) level is measured by NEXTCLINICS Czech a.s. The reference range is 3,30-5,59 mmol/l.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Pavel Kolar´s Centre of Physical Medicine, Prague
  - The Faculty of Physical Education and Sport, Charles University, Prague

IPD SHARING:
Plan to Share IPD: No
Due to the sensitivity of the data (personal data), it has not been decided whether the data will be provided to third parties.

REFERENCES:
- [Derived] Jurik R, Stastny P, Kolinger D, Gola A, Vetrovsky T. Blood pressure changes during different methods of resistance training in normotensive and stage 1 hypertensive individuals: a repeated measures cross-sectional study. BMC Sports Sci Med Rehabil. 2025 Mar 14;17(1):49. doi: 10.1186/s13102-025-01097-3. PMID 40087719